CLINICAL TRIAL: NCT05487105
Title: Addendum Elternwerden in Zeiten Der COVID-19-Pandemie Zum Projekt "Pränatales Lernen Und Wiedererkennen Von Auditiven Reizen - Eine Psychophysiologische Perinatal Studie"
Brief Title: Becoming a Parent During the COVID-19 Pandemic in Austria and Germany
Status: Completed | Type: Observational
Sponsor: University of Salzburg (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Cristina Florea, Prinicipal Investigator, University of Salzburg
Other Study IDs: EK-GZ12/2013-Addendum-07/2021
Record Dates: First submitted 2022-07-29; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Parents; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an online survey in Austria and Germany directed at parents with children born since the start of the first lockdown of the COVID-19 pandemic (birthdate beginning with 16.03.2020). The survey includes questions about:

* current stress levels and depressive symptoms,
* resilience during the pandemic,
* social support,
* retrospective birth risk factors, pregnancy distress and pregnancy experience,
* demographic factors and
* other questions related to parenting and the COVID-19 pandemic.

DETAILED DESCRIPTION:
The study evaluated data collected in the course of an online survey during the COVID-19 pandemic in Austria and Germany. The questions were conceived to reflect aspects of pregnancy, childbirth and early child rearing that could be affected by the pandemic, and included commonly used and previously validated scores for assessing pregnancy distress (Pregnancy Distress Questionnaire, PDQ), birth experiences (Childbirth Experience Questionnaire 2, CEQ2) postnatal depression (Edinburgh Postnatal Depression Scale, EPDS), perceived stress (Perceived Stress Scale, PSS) and pandemic-related experiences (pandemic resilience part, adapted to postnatal period, from the Pandemic Related Stress in Pregnancy Scale, PREPS). In addition, the investigators composed questions and scales that referred to specific pandemic- and parenting-related issues that were not covered otherwise. The investigators also tried to question both the fathers and the mothers, and consequently mothers received more pregnancy-related questions than fathers. Furthermore, biological mothers received childbirth-related questions which were omitted for adoptive mothers.

ELIGIBILITY:
Inclusion Criteria:

* parents that had a baby born since the 16th of March 2020 (which corresponds to the beginning of the first lockdown in Austria and in Bavaria, Germany)
* living in Austria or Germany

Exclusion Criteria:

* stillborn or neonatal death

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents that had a baby born since the 16th of March 2020 (which corresponds to the beginning of the first lockdown in Austria and in Bavaria, Germany)
Sampling Method: Non-Probability Sample
Enrollment: 2226 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Over the previous seven days from the time of answering the questionnaire
  Score on the Edinburgh Postnatal Depression Scale, range 0-30. Interpretation: 0-8 (depression not likely), 9-11 (depression possible), 12-13 (fairly high possibility), 14-30 (probable depression).
Perceived stress | Over the previous month from the time of answering the questionnaire
  Score on the Perceived Stress Scale, range 0 to 40. Interpretation: 0-13 (low stress), 14-26 (moderate stress), 27-40 (high stress).
Childbirth experience | At 0 to up to 15 months after birth (one assessment)
  Score on the Childbirth Experience Questionnaire 2 - factors "Coping ability", "Participation" and "Emotional experience". Range 13 (negative) to 52 (positive birth experience).
Pregnancy distress | At 0 to up to 15 months after birth (one assessment)
  Score on the Pregnancy Distress Questionnaire, 10 items scored from 0 to 4. The total score is the sum of all items divided by the number of items (10). The score's range is 0 (low distress) to 4 (high distress).
Resilience during the pandemic | One year after the beginning of the COVID-19 pandemic
  Score on the resilience subscale from the Pandemic Related Pregnancy Stress Scale, adapted to postpartum participants. It contains 7 items, scored from 1 to 5. The total score range is 7 (low resilience) to 35 (high resilience).
Social support | At 0 to up to 15 months after birth (one assessment)
  The Social Support score consisted of 3 Items scored on a Likert scale from 0-4, covering the subjective feeling of social support. Its possible range was 0 to 12, with higher scores indicating more social support.
Child's Social Contacts | At 0 to up to 15 months after birth (one assessment)
  The Child's Social Contacts score is the sum of frequencies with which the child has contact with other people, each item representing one person/relationship (mother, father, siblings, grandparents, other adults, other children), which are independent of each other. The possible range for the Child's Social Contacts score was 0-6, 6 points indicating daily contact with parents, sibling(s), grandparent(s), other adults, and other children, and 0 indicating no contact at all.
Pandemic Repercussions | One year after the beginning of the COVID-19 pandemic
  The Pandemic Repercussions score comprises five items which inquire about the perceived influence of the coronavirus situation on the pregnancy, birth experience, health and development of the child, financial security, and on the partnership. Each item was scored from -2 (for strong positive influence) to 2 (strong negative influence), making the possible range of the score from -10 to +10, where negative values indicate positive repercussions and positive values indicate negative repercussions.
Pandemic Distress | One year after the beginning of the COVID-19 pandemic
  The Pandemic Distress score consisted of 3 Items that inquired about the participant's worries about the virus affecting herself, her relatives and/or her baby. Each item was scored on a Likert scale from 0-4, so that the possible range of the score was 0-12, with higher values indicating that the participant is more worried. This score is computed only for those participants who had not had Covid-19 themselves, since those who had had Covid-19 were not asked whether they worried to catch it again.
Birth Risk | Retrospectively assessed, at 0 to up to 15 months after birth (one assessment).
  The Birth Risk score consists of 10 items which reflect the medical risk factors for a poor birth outcome: whether singleton or multiples pregnancy, pre/at/post-term birth, newborn weight at birth, type of birth, maternal age, quarantine during birth, history of miscarriage, mother's parity (higher risk if first or fifth/further pregnancy), length of hospitalization for the mother and for the baby. This score had a possible range of 5 to 29, with lower values indicating smaller risk and higher values higher risk.

SECONDARY OUTCOMES:
Correlations between the scores from the primary outcome measures | At the time of answering the questionnaire
  Spearman correlations between the scores from the primary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Schabus, Prof. Dr., Study Chair — Paris-Lodron University of Salzburg; Monika Angerer, Dr., Principal Investigator — Paris-Lodron University of Salzburg
Locations (1):
- Paris-Lodron University of Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: Yes
The anonymously collected data including the answers to the questionnaire, the questionnaire itself, and the analytic code shall be shared on an open data platform at the end of the study.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The data will be uploaded by December 2022 and will be available for an unlimited time.
Access Criteria: Researchers from accredited institutions.
URL: https://aussda.at/en/